CLINICAL TRIAL: NCT05065060
Title: Parkinson's Progression Markers Initiative Online Study (PPMI Online)
Brief Title: Parkinson Progression Marker Initiative Online (PPMI Online)
Status: Recruiting | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Caroline M Tanner, Protocol Co- Principal Investigator, University of California, San Francisco
Other Study IDs: PPMI-007
Record Dates: First submitted 2021-09-02; First posted 2021-10-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Neurodegenerative Disorder; Prodromal; At Risk; Participant Reported Outcomes
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
Parkinson Progression Marker Initiative Online (PPMI Online) is an observational study collecting participant reported information from people with and without Parkinson's disease (PD), for the goal of better understanding risk and predictive factors for PD.

PPMI Online is part of the broader Parkinson Progression Marker Initiative aimed at identifying markers of disease progression for use in clinical trials of therapies to reduce progression of PD disability.

DETAILED DESCRIPTION:
PPMI is a broad program that is expanding the goals of the original PPMI study, and will include this PPMI Online protocol, as well the PPMI Clinical [NCT04477785], PPMI Remote, PPMI Digital protocols (with external regulatory oversight). All participants in PPMI may be asked to participate in one or all of these protocols and their enrollment in these studies may occur in varying order. PPMI participants may also be asked to participate in additional PPMI companion studies (as they are developed), which may only involve a subset of PPMI participants based on their cohort designation

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Disease (PD) Participants:

  * Male or female age 18 years or older.
  * Has received a diagnosis of Parkinson's disease

Participants without PD:

* Male or female age 18 years or older.
* Has not received a diagnosis of Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In PPMI Online, up to 500,000 participants with and without PD will be enrolled and contribute data longitudinally and cross-sectionally using a web-based platform.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2041-12 (Estimated); Study Completion 2041-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Ib & II | Baseline to 240 months
  Evaluates self-reported motor and nonmotor Parkinson's disease symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tanner, MD, PhD, Principal Investigator — University of California, San Francisco; Kenneth L Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- UCSF Movement Disorders and Neuromodulation Center (MDNC), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pierz KA, Aamodt W, Gochanour C, Kurth R, Brumm MC, Coffey CS, Heathers LE, Totten M, Doty RL, Marek K, Siderowf A; Parkinson's Progression Markers Initiative. Percentile scores for the revised University of Pennsylvania Smell Identification Test for 16,972 individuals 60 years of age and older. NPJ Parkinsons Dis. 2025 Oct 1;11(1):280. doi: 10.1038/s41531-025-01095-9. PMID 41034300